CLINICAL TRIAL: NCT01282554
Title: Evaluation of Electrostimulation Program During Dialysis Sessions in Chronic Renal Failure Patients
Acronym: EMS-Dialyse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-A01149-30
Record Dates: First submitted 2010-12-30; First posted 2011-01-25 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Chronic Renal Failure (CRF)
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- stimulated group (Experimental): stimulated group
  Interventions: Device: electrostimulation program (Rehab 400)
- control group (No Intervention): Control group : non stimulated group.

INTERVENTIONS:
Device: electrostimulation program (Rehab 400) — electrostimulation program (Rehab 400) : electrostimulation program during dialysis sessions for 3 months.
  Electrostimulation modalities have been chosen to seek both slow and fast muscle fibers : 35 Hz ; impulsion time: 400 µsec ; on/ off : 7'' contraction / 8'' relaxation. Stimulated muscles are quadriceps. Electrostimulation time will be 30 minutes. Each patient will individually regulate work intensity, maximal intensity should be the maximal tolerable intensity.
  Electrostimulation will be done 3 times per week. In case of asthenia or medical condition, electrostimulation can be delayed. The program will take place for 3 months.
  Other Names: electrostimulation
  Arms: stimulated group

SUMMARY:
Sport improves quality of life and health, decreasing cardiovascular risks and increasing effort tolerance. Chronic renal failure (CRF) induces many clinical and biological complications leading to less effort tolerance (strength and endurance). Renal failure patients got also many cardiovascular risks : sedentarily lifestyle, hypertension (HTA), diabetes, neuropathies, bone disorders, depression and sedentarity due to dialysis sessions. Moreover, dialysis sessions three times a week induce the spiral of deconditioning. In order to counteract this, sport should be encourage in this specific hemodialysis population.

The aim of this study is to evaluate electrostimulation program during dialysis sessions for 3 months. Evaluation will be done using the Test of 6-minute walk (6MWT).

Secondary aims will be evaluated:

* Muscular strength and quadriceps diameter
* Equilibrium
* Quality of life.
* Strength developed during maximal exercise test in a subgroup (patient undergoing dialysis in Rennes center, about 40% of the total population)
* Nutritional intakes (quantitative and qualitative evaluation)

DETAILED DESCRIPTION:
The primary outcome is the difference between distances during the 6 minutes walk test before and after the 3 month program between the stimulated and the non stimulated group.

The secondary outcomes will be evaluated by maximum strength developed during the ergometry, limited by symptoms; maximal charge during muscular test; quadricipital diameter; time for the " Timed up and go " test; quality of life scores. All those scores will be evaluated in the control and stimulated groups before and after the 3 month period.

This is an open randomized controlled study. Tests will be done by an investigator unaware of the stimulation group. The study is designed to detect a difference of 61 m (+/- 80 m) (6MWT) before and after stimulation in the stimulated group and 0 in the control group. This difference has been based on a pilot study with ergocycle in the same population and on literature in other populations (chronic respiratory failure or post cardiac surgery). We estimated that 70 patients would need to be enrolled in each group to provide 90% statistical power with a bilateral test.

ELIGIBILITY:
Inclusion Criteria:

* Patients, > 18 y/o, undergoing chronic hemodialysis since more than 3 months.
* Physical activity score (Voorrips test) <9.4
* Patients clinically and hemodynamically stable.
* No major drug or dialysis treatment changes since 2 weeks
* Written consent signed.

Exclusion Criteria:

* Relative or absolute contraindication to ergotest (ACC/AHA, 2002) and/or physical reentrainment.
* Incapacity to practice the Test of 6-minute walk (6MWT) or ergotest
* Clinical instability during hemodialysis sessions.
* Hb<9g/dl despite medical treatment ; PAS ≥180 mmHg et/ou PAD ≥110 mmHg despite medical treatment ;
* Cardiac pace maker or defibrillator ;
* Pregnancy ;
* Recent cardiovascular events: cardiac failure less than 10 days before, instable angina, coronary angioplasty less than 10 days cardiac surgery less than 1 month, valvulopathy requiring surgery, myopericarditis, severe Rhythm troubles despite medical treatment, stade IV arteriopathy.
* BMI ≥ 30 kg/m² ;
* Anxiety and mental disorder
* Concomitant pathology leading to severe general status alteration.
* Patient participating to another medical study
* Electromyostimulation or effort entrainment program less than a month.
* Patients on renal transplantation awaiting list.
* Patient practicing sport ( response to Voorips test)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
difference between distances during the 6 minutes walk test before and after the 3 month program between the stimulated and the non stimulated group | 3 months
  The primary outcome is the difference between distances during the 6 minutes walk test before and after the 3 month program between the stimulated and the non stimulated group

SECONDARY OUTCOMES:
maximum strength developed during the ergometry, limited by symptoms; maximal charge during muscular test; quadricipital diameter; time for the " Timed up and go " test; quality of life scores. | 3 months
  The secondary outcomes will be evaluated by maximum strength developed during the ergometry, limited by symptoms; maximal charge during muscular test; quadricipital diameter; time for the " Timed up and go " test; quality of life scores. All those scores will be evaluated in the control and stimulated groups before and after the 3 month period.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Laruelle, MD, Principal Investigator — Rennes University Hospital
Locations (11):
- France (11):
  - AUB Santé Brest, Brest, Brittany Region
  - AUB Santé Fougères, Fougères, Brittany Region
  - AUB Santé Lorient, Lorient, Brittany Region
  - AUB Santé Montgermont, Montgermont, Brittany Region
  - AUB Santé Morlaix, Morlaix, Brittany Region
  - AUB Santé Quimper, Quimper, Brittany Region
  - Rennes University Hospital, Rennes, Brittany Region
  - AUB Santé Rennes, Rennes, Brittany Region
  - Cholet Hospital, Cholet
  - Nantes University Hospital, Nantes
  - ECHO Nantes, Nantes

REFERENCES:
- [Result] Besnier F, Laruelle E, Genestier S, Gie S, Vigneau C, Carre F. [Effects of exercise training on ergocycle during hemodialysis in patients with end stage renal disease: relevance of the anaerobic threshold intensity]. Nephrol Ther. 2012 Jul;8(4):231-7. doi: 10.1016/j.nephro.2011.10.002. Epub 2011 Nov 18. French. PMID 22100992